CLINICAL TRIAL: NCT04703062
Title: The Effects of Exercise Training on Physical Activity Level, Daily Living Activities and Participation in Children With Hemophilia
Brief Title: The Effects of Exercise Training in Children With Hemophilia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Canan Atay, principal investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 13022260-300-63450
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Hemophilia
Keywords: hemophilia; exercise; participation; physical activity; muscle strength
MeSH Terms: conditions — Hemophilia A; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group 1 (Experimental): physical activity counseling group + exercise group
  Interventions: Behavioral: Experimental group 1
- Experimental group 2 (Experimental): physical activity counseling group
  Interventions: Behavioral: Experimental group 2

INTERVENTIONS:
Behavioral: Experimental group 1 — It is planned to do exercises for 50 minutes a day, 2 days a week during 8 weeks with physiotherapist. It will be planned individually according to the needs of the patients. Exercises will progress in the following weeks by changing the number of repetitions, the amount of resistance and the amount of time. Counseling about physical activity and the suggested sports activity will be provided. In daily living activities ergonomics and joint protection principles will be taught. Informing Family.
  Other Names: exercise
  Arms: Experimental group 1
Behavioral: Experimental group 2 — Counseling about physical activity and the suggested sports activity will be provided.Patients make aerobic and strengthening exercises by himself based on physiotherapist's suggestions. Informing Family about; Why are the exercises necessary To what extent the families should be protective The harmful effects of inactivity There will be information about the resting-activity cycle when there is bleeding.
  Arms: Experimental group 2

SUMMARY:
This study aims to investigate the effects of an individually planned exercise program, counseling and family education on the followings in patients with hemophilia (PWH);

1. To examine the joint range of motion, muscle strength and functional status.
2. To evaluate the level of physical activity and daily living activities
3. To aim to determine the amount of change after participation.

DETAILED DESCRIPTION:
Hemophilia is defined as bleeding in the musculoskeletal system and soft tissues as a result of the lack of clotting factors in the blood. Recurrent attacks of hemarthrosis cause pain, also because of the pain patients tend to use joints less than usual. The decrease in joint movement makes it harder to return to active movement again. There is a limited literature on the effects of exercise on children with hemophilia.

Hemophilia is a hereditary bleeding disorder that develops as a result of factor VIII or IX deficiency; it is a rarely seen disease that discloses itself by hemarthrosis and intramuscular bleeding. Factor VIII deficiency is called Hemophilia A and Factor IX deficiency is called Hemophilia B. This disease is inherited by the X chromosome and passes on to male children through female carriers. Although Hemophilia A is observed rarely, one in about 5,000-10,000 male births, its frequency is still 5-6 times higher than Hemophilia B. Around 70% of hemophilia A patients have more severe disease, however, this rate is approximately 50% in hemophilia B.

Hemophilia patients experience bleeding in the musculoskeletal system and soft tissues as a result of the lack of clotting factors in the blood. Recurrent attacks of hemarthrosis cause pain, also because of the pain patients tend to use joints less than usual. Decrease in joint movement makes it harder to return to active movement again in the majority of the cases, bleeding occurs into the joint (mostly the knee, elbow and ankle) and only a small part of the bleedings occurs into the muscle (especially the iliopsoas, calf and forearm muscles).

In order to be able to participate according to the international classification of functions of health (ICF), it is prioritized that the activities are functional.

Targeted treatment is a functional treatment application that conforms to ICF's "activities and participation among children. An activity is carrying out of a task or movement by an individual and the difficulties faced while carrying out the tasks or movements is called limitations. Participation means the individual's being in life. In life conditions, problems confronted are participation restrictions. Activity limitations can often lead to participation restrictions.

Fear of bleeding in pediatric patients, particularly from the period of childbirth leads families to form an immobile lifestyle for their children compared to healthy individuals.

The recurrent bleeding often occurs in the lower extremity joints, it causes pain and swelling, therefore patients need to keep the joint immobile which is particularly the reason why patients spend these periods mostly resting. So then, again, patients forfeit activity for fear of recurrent bleeding. The decrease in activity leads to a loss of strength and balance. Also, sports that could lead to bleeding or trauma are not suitable for hemophilia patients. The benefits and risks of sports activities for hemophilic individuals should be well known and the patient should be oriented toward suitable sports. For this reason the rehabilitation program should be arranged as a personalized and systematic program according to local and general joint and muscle conditions.

Hematologic therapy alone is not sufficient for the treatment of musculoskeletal bleeding. The sedentary lifestyle that develops with hemophilic arthropathy often leads to immobility problems such as decreased muscle strength, weak balance and coordination, increased risk of obesity. These problems lead to instability and changes in joint loads, thereby instances of new bleeding and increased joint damages. In a similar way, after hemarthrosis, in acute situations, if the necessary period of resting is not accompanied by an appropriate physiotherapy, it causes a vicious cycle of immobility, new bleeding and eventually hemophilic arthropathy and loss of function.

The key to the successful management of hemophilic arthropathy is to begin the treatment early. The first step of treatment for hemophilic arthropathy is physiotherapy with factor replacement to prevent bleeding attacks and joint damage before hemarthrosis progresses to chronic synovitis and joint erosion.

Physical activity means body movement by using energy and exercise means planned physical activities that are personally structured. Regular exercise can prevent the progression of hemophilic arthropathy or it may reduce the risk. Therapeutic exercises are the main elements of rehabilitation for Patients with hemophilic arthropathy and muscle bleeding.

The main objective of therapy should be the following: restoration or preservation of range of motion, strengthening of muscles, prevention or treatment of joint contracture, pain management, increasing exercise tolerance, improvement of balance, coordination, and proprioception. To prevent patients from giving up on exercising earlier than required, İt is important to assist patients, encourage them during exercises, support them and when necessary give them advice and explain the exercises in a way that patients can easily and clearly understand. There is a fine line between beneficial and harmful activities, this fine line leads many patients with bleeding disorder to avoid exercise for fear of causing bleeding. Paradoxically, when people with bleeding disorders avoid exercising this causes decreased function, range of motion, and quality of life because of muscle weakness.

In Turkey, the cost of joint health complications in patients with hemophilia and other inherited bleeding disorders is significantly high however most significant point is that these costs can be avoided. Physical activity which is a non-pharmacologic treatment method, plays an important role in reducing the risks, alleviating the symptoms and improving the results in hemophilia. For this reason, it is very important to develop strategies to increase the level of physical activity.

In the relevant literature there are very few studies on the effects of exercise in pediatric patients with hemophilia. With this study, we plan to show, in an objective manner, that the personally planned exercise program leads to change in the level of physical activity, activities of daily life and participation.

The Methods of the Study

Before the study the patients and their families will be informed about the evaluations, treatments that will be made. They will be also informed about outcomes and evaluations after the treatment, and the risks that they may face during the the treatments. They will also be asked to sign the "Informed Consent Form" for their voluntary participation in the study.

An "Assessment Form" will be prepared in order to keep the record of demographic and disease information of all the cases included in the study. Hemophilia types, patients biographic information, family history, the time when the disease was diagnosed, treatments taken, medications used, body mass index, range of motion and muscle strength will be recorded in this assessment form.

Randomly patients will be divided into two groups as physical activity counseling and individually planned exercise group and only physical activity counseling group. We plan that the exercise will be done for 50 minutes a day, twice in a week and will last for 8 weeks.

Before and after the 8-week intervention program of all patients physical activity levels with International Physical Activity Questionnaire (IPAQ), activity performance exercise with Children's Functional Independence Scale (Wee-FIM) and Canadian Occupational Performance Measurement (COPM), joint health with hemophilia joint health scoring (HESS), exercise capacity with 6-minute walking test (6MWT) and sit-and-stand test, hand function speed and dexterity with Jebsen-Taylor Hand Function Test (JTHFT) and quality of life with Pediatric's Quality of life Scale (PedsQL) will be evaluated.

Assessment methods, exercise and counseling practices will be carried out in the Turkey Hemophilia Society of Physiotherapy Unit.Only the participants in the hematologists follow-up will continue their routine doctor checks and recommendations.

All analyzes will be performed using Statistical Package for Social Sciences (SPSS) for Windows 22. The compliance of the data to normal distribution will be evaluated by drawing the Kolmogorov-Smirnov test and histogram. Parametric tests will be used for data suitable for normal distribution. Data that are not suitable for normal distribution will be analyzed with non-parametric tests. Variables will be defined by their mean and standard deviation values. Analyzes and correlations between groups will be examined separately with appropriate tests. A value of p<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Being in the 7-18 age range
* Being diagnosed with hemophilia A or B
* Having an ongoing prophylactic treatment
* Having a heavy or middle Factor level
* Volunteering to exercise at 2 days a week in the intervention group within the scope of the research
* Being able to communicate in Turkish written and verbal

Exclusion Criteria:

* Being in period of active bleeding
* Having Body mass index over 30 kg / m²
* Having an additional neurological diagnosis that will influence work and cooperation

Ages: 8 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
Hemophilia Joint Health Scoring (HJHS) | through study completion, an average of 1 day
  Because hemophilic individuals have a high risk of arthropathy, joints with bleeding should be examined very closely and arthropathic diagnosis should be detected at an early stage. For this reason, the HJHS was developed by the Physiotherapy Subgroup of the International Prophylaxis Working Group, this groups is made up of expert physiotherapists, rheumatologists and hematologists. It has been stated that HJHS is more sensitive than X-ray in diagnosing arthropathy findings, and it is used for about 40-60 minutes. Also, it has been reported that MRI and ultrasonography are not sufficient in joint evaluation when they are used alone; It has been shown that it should be performed together with HESS. The maximum disease score for each joint is 20, with a possible total score of 120, plus a maximum of four for global gait. High score means worse joint health.
BMI (body mass index) | through study completion, an average of 1 day
  Weight and height will be combined to report BMI in kg/m^2. Underweight = <18.5 Normal weight = 18.5-24.9 Overweight = 25-29.9. Obesity = BMI of 30 or greater
Canadian Occupational Performance Measurement (COPM) | through study completion, an average of 1 day
  An individual-oriented self-assessment report in the COPM will be used to test participation restrictions. An increase in performance and satisfaction score means that the patient has improved his/her performance in doing the activity and that he/she has an increased satisfaction over this performance. It is a generic measure suitable for all clients with perceived problems in daily activities. The COPM results in two scores (performance and satisfaction) each of 10. The patient prioritizes up to five problems she/he deems are the most urgent or important and rates the problems on an ordinary 10-point scale regarding performance (1=not able to do at all and 10=able to do extremely well) and satisfaction (1=not satisfied at all and 10=extremely satisfied). Performance and satisfaction scores for the top 5 activities were summed and divided by the number of activities, resulting in total performance and satisfaction scores.
range of motion (ROM) | through study completion, an average of 1 day
  Elbow, knee and ankle flexion and extension active ROM are measured using a universal goniometer. In this study, 3 repetitions are performed in each direction, and the average value is recorded for analysis. Interrater reliability of measurements of ROM for upper extremity joints were ICC = 0.75.15
muscle strength | through study completion, an average of 1 day
  The muscle strength of elbow, knee and ankle flexor and extensors are measured using a hand-held dynamometer (The Lafayette Instrument Company). The measurements are recorded in kg/N. This dynamometer allowed a measurement of muscle strength from 0.0 to 199.9 kg, with 0.1 kg precision.
  The test participants are asked to forcibly contract their muscle while a resistive force is applied by the dynamometer in the opposite direction of the intended movement. During the test, the device recorded the maximal isometric strength of the muscle in kg/N. Each muscle is assessed 3 times, and the mean value is calculated. Test-retest reliability in hand-held dynamometry in children has been reported, and test-retest correlation coefficients ranged from 0.74 to 0.99 in their study.
The Pediatric's Quality of life Scale (PedsQL) | through study completion, an average of 1 day
  PedsQL will be evaluated with the quality of life for children scale. The parent form will be filled by the person two takes care of the child and the child from will be filled by the child who participated to the study these forms will be filled separately and simultaneously. Scoring will be made in 3 areas. First of all the overall score of the scale will be calculated, second the physical health score will be calculated and third the psychosocial health total score which consists of emotional, social and school functionality scores will be calculate. The scale consists of child self-report and parent proxy reports. The scale includes a total of 23 items. The total scale score, physical health summary score, and psychosocial health summary score were calculated. Items were scored between 0 and 100: 0 (100) = never a problem; 1 = (75) almost never; 2 = (50) sometimes; 3 = (25) almost always; and 4 = (0) always. Higher PedsQL scores indicate better HRQoL.

SECONDARY OUTCOMES:
Long version of International Physical Activity Questionnaire (IPAQ) | through study completion, an average of 1 day
  Long version of IPAQ will be used to measure physical activity level. There are three levels of physical activity proposed to classify populations - 'low', 'moderate', and 'high' Vigorous Intensity = 8.0 metabolic equivalent (METs) Moderate Intensity = 4.0 METs. Low Intensity = 3.3 METs
6 minutes walk test | through study completion, an average of 1 day
  6 minutes walk test will be used to measure exercise capacity The six minute walk distance in healthy adults has been reported to range from 400m to 700m Age and sex-specific reference standards are available and may be helpful for interpreting 6MWT scores for both healthy adults and those with chronic diseases 47 . However, it is difficult to use normative values because of the differing methods used in studies. An improvement of 54m has been shown to be a clinically important difference24 in a study of people with chronic lung disease which is similar to the recommended criteria of meaningful clinical change of 50m based on analyses from a sample of 692 community living older adults and individuals who have survived a stroke 25.
Children's Functional Independence Scale (Wee-FIM) | through study completion, an average of 1 day
  "Children's Functional Independence Scale (Wee-FIM)" will be used to determine the problems related to activity performance. In total, Wee-FIM consists of 6 areas including sphincter control, self-care, communication, locomotion, social-cognitive and transfers. For each of item in these sections, a score of 1 to 7 is used to evaluate whether or not the patient performs the function on time, whether or not he/she receives assistance, or needs an auxiliary device. A participant can get a minimum of 18 (fully dependent) or a maximum of 126 (fully independent).
Sit-and-Stand Test | through study completion, an average of 1 day
  With a "Sit-and-Stand Test" , the participant who sits in a 43 cm high standard chair with his arms crossed on his shoulders, is asked to stand up and sit quickly for 30 seconds and the number of times that teh stand up position is achieved is recorded.
Jebsen Taylor Hand Function Test | through study completion, an average of 1 day
  Hand function speed and dexterity were assessed with the JTHFT, which is a commonly used standardized test for assessing upper extremity efficiency; it is reliable, valid and normative for children. The jebsen test evaluates both the dominant and nondominant hand skills and supplies an objective assessment of the hand function involved in a series of 7 subtests of activities of daily living (ADL). We used the subtests of writing; turning over cards; picking up a small common object; stacking checkers; simulated feeding; (6) moving light and heavy objects on a board. The time (in seconds) taken to perform the 7 subtests was measured with the same stopwatch. The writing subtest was conducted, assessed, and scored with only the dominant hand. The reliability of the JTHFT for children has previously been reported (the dominant and nondominant hands were intraclass correlation coefficient (ICC) 0.74 and 0.72, respectively)

CONTACTS AND LOCATIONS:
Overall Officials: Ela Tarakcı, prof dr, Study Chair — Istanbul University- Cerrahpasa Physiotherapy and Rehabilitation Department
Locations (1):
- Canan Atay, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: An institutional pilot study to investigate physical activity patterns in boys with haemophilia — https://pubmed.ncbi.nlm.nih.gov/27530715/
- See also: Physical exercise, pain and musculoskeletal function in patients with haemophilia — https://pubmed.ncbi.nlm.nih.gov/27075748/
- See also: Effects of a 6-week, individualized, supervised exercise program for people with bleeding disorders and hemophilic arthritis — https://pubmed.ncbi.nlm.nih.gov/20203091/
- See also: Exercise may decrease further destruction in the adult haemophilic joint. — https://pubmed.ncbi.nlm.nih.gov/16643207/
- See also: Guidelines for the management of hemophilia — https://pubmed.ncbi.nlm.nih.gov/22776238/